CLINICAL TRIAL: NCT04383717
Title: The Efficacy of Levamisole and Isoprinosine in the Treatment of COVID19: A Proposed Therapeutic Trial
Brief Title: Levamisole and Isoprinosine in the Treatment of COVID19: A Proposed Therapeutic Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dermatology Lecturer Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Levamisole and isoprinosine
Record Dates: First submitted 2020-05-04; First posted 2020-05-12 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Tract Infections
Keywords: Levamisole; Isoprinosine; COVID19
MeSH Terms: conditions — Respiratory Tract Infections; COVID-19 | interventions — Levamisole; Inosine Pranobex; Azithromycin; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proposed treatment group (Active Comparator): Levamisole and isoprinosine
  Interventions: Drug: Levamisole and isoprinosine
- Control group (Active Comparator): hydroxychloroquine and azithromycin
  Interventions: Drug: Azithromycin and hydroxychloroquine

INTERVENTIONS:
Drug: Levamisole and isoprinosine — oral tablets levamisole 50 mg 3 times daily every other day for 2 weeks Isoprinosine oral tablets 1 g 4 times daily for 2 weeks
  Other Names: ketrax and inosiplex
  Arms: Proposed treatment group
Drug: Azithromycin and hydroxychloroquine — oral tablets daily 500 mg azithromycin Oral tablets daily 200 mg hydroxychloroquine twice daily
  Other Names: Zithromax and plaquinel
  Arms: Control group

SUMMARY:
The use of both levamisole & Isoprinosine has both synergistic and complementary effect in the treatment of COVID 19 infection

DETAILED DESCRIPTION:
Study design: Randomized controlled trial, randomization by closed envelope technique Informed consent will be written for each patient of either group

At the beginning of the study all patients will have the following investigations done: CBC with differential, ESR, PCR for COVID 19, D dimer and CT chest and confirmed cases will included in the study

Pregnant and lactating women together with children with other comorbidities will be excluded from the study

Study groups:

Duration of the study is 4 weeks

Both groups with persistent COVID 19 symptoms that require hospitalization

Group 1: 30 patients with confirmed COVID19 infection and sharing clinical features like fever, malaise, sore throat, runny nose, persistent cough &dyspnea, requiring hospitalization

Group 2: control group: 30 patients

Treatment endpoint • Cure of patients: Improvement of symptoms Laboratory findings ESR and total leucocytic count returning to normal PCR negative Radiological improvement

• Worsening of symptoms or fatalities

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID 19 infection (positive PCR, elevated ESR, leucopenia)
* Clinical picture of COVID 19 infection including fever, malaise, sore throat, coughing, dyspnea, and runny nose

Exclusion Criteria:

* Mild cases of COVID 19 that do not require hospitalization
* Pregnant & lactating women
* Children with other comorbidities
* People who received previous treatment for COVID 19 in the last 2 weeks N.B. Diabetes and hypertension not excluded

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-05 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
COVID 19 induced fever in both groups | 4 weeks
  Improvement of fever in degrees celsius
COVID 19 induced dyspnea in both groups | 4 weeks
  improvement of dyspnea by normalization of respiratory rate
COVID 19 viral load in both groups | 4 weeks
  PCR of COVID 19 changes from positive to negative

SECONDARY OUTCOMES:
laboratory clearance in both groups: CRP in mg/dL | 4 weeks
  CRP in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El Darouti, Professor, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No